CLINICAL TRIAL: NCT05846438
Title: Effect of Drain Care on Infection Rate and Quality of Life in Implant-Based Breast Reconstruction.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Stephen Colbert, Division Chief of Plastic and Reconstructive Surgery, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2092673
Record Dates: First submitted 2023-04-05; First posted 2023-05-06 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Infections; Quality of Life
MeSH Terms: conditions — Infections | interventions — Postoperative Period

STUDY DESIGN:
Intervention Model Description: The investigators have two groups of patients. Group one will be allowed to shower 48 hours after surgery. Group two will not be allowed to shower until the drains are removed.
Masking Description: The study is unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Showering 48 hours after Surgery (Experimental): Group 1 will be allowed to shower 48 hours after surgery with drain tubes still in place.
  Interventions: Other: Showering 48 hours after surgery
- Showering after drain tubes are removed (No Intervention): Group 2 will not be allowed to shower until drain tubes are removed.

INTERVENTIONS:
Other: Showering 48 hours after surgery — The main intervention is allowing patients to shower 48 hours after surgery
  Arms: Showering 48 hours after Surgery

SUMMARY:
The goal of this clinical trial is to learn whether showering with surgical drain tubes in place after first stage breast reconstruction causes increased risk of infection. The main questions it aims to answer are:

* Is there an increased risk of infection/complications with showering 48 hours after drain tubes are in place
* Does showering after 48 hours with drain tubes in place affect quality of life.

DETAILED DESCRIPTION:
SSI (soft tissue infection) is an aggravating risk specifically associated with implants. Breast reconstruction quotes infection rates anywhere from 1-35% while cosmetic augmentations quote rates around 1.5%. Usually, the causative organisms are skin flora like Staph aureus and Staph epidermidis. Occasionally mycobacterium and other atypical bacterium are isolated more commonly in the immunocompromised. Despite perioperative antibiotics, SSI is still a prevalent complication increasing total expenditure of patients and hospital systems upwards of $4000/patient in reoperation fees and hospital stay costs. Skin prep and antibiotics in the preoperative phase is very important to the sterile technique and decreasing risk of infection by decreasing bacterial load at the time of incision and surgery. However, postoperative care and interventions are less strictly evaluated and defined. Currently, there is no standard of care in regards to showering post operatively with JP (Jackson-Pratt) drains in place. Timing of showering is ultimately based on surgeon preference. In practice, the investigators routinely have had patients wait to shower until the JP drains are removed. The investigators hypothesize that showering daily, even with drains in place, will not increase rates of infection in breast reconstruction and perhaps improve quality of life during first stage. This study is prospective with participants randomized to either shower daily after 48hrs or standard of care and shower after drains removed. The participants will be asked to fill out a quality of life survey 90 days after enrollment. The patients will also be monitored for signs of infection for 90 days.

ELIGIBILITY:
Inclusion Criteria:

* undergoing breast surgery with placement of tissue expander and drains, acceptance of protocol and procedures, age > 18

Exclusion Criteria:

* no existing wounds, previous infections related to implant device if delayed, refusal by patient

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The study will involved patient's undergoing breast reconstruction following mastectomy.
Enrollment: 100 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Presence of Post Operative Infection | 90 days
  The primary outcome measure will be the presence of infection as judged by the non blinded attending surgeon within the 90 day time frame during post operative evaluations. A breast infection is defined as increased erythema, warmth, and pain at the breast or systemic symptoms such as fevers and chills. Breast infections will be treated with a course of IV antibiotics and possible tissue expander removal and breast pocket irrigation and debridement in the operating room. If the attending physician determines that an infection is present any time during the treatment period the patient will be categorized as infected.

SECONDARY OUTCOMES:
Quality of Life Survey | 90 days
  Subjects will complete a survey at 90 days using a scale from 0 (strongly disagree) to 5 (strongly agree) indicating how showering or not showering with drain tubes in place affected their quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ogawa H, Tahara S. Postoperative Showering for Patients With Closed Suction Drainage: A Retrospective Cohort Study of Deep Inferior Epigastric Perforator Flap Breast Reconstructions. Cureus. 2022 Mar 30;14(3):e23665. doi: 10.7759/cureus.23665. eCollection 2022 Mar. PMID 35505721
- [Background] Gowda AU, Chopra K, Brown EN, Slezak S, Rasko Y. Preventing Breast Implant Contamination in Breast Reconstruction: A National Survey of Current Practice. Ann Plast Surg. 2017 Feb;78(2):153-156. doi: 10.1097/SAP.0000000000000822. PMID 27464530
- [Background] Elder EE, Brandberg Y, Bjorklund T, Rylander R, Lagergren J, Jurell G, Wickman M, Sandelin K. Quality of life and patient satisfaction in breast cancer patients after immediate breast reconstruction: a prospective study. Breast. 2005 Jun;14(3):201-8. doi: 10.1016/j.breast.2004.10.008. PMID 15927829
- [Background] Hanna KR, Tilt A, Holland M, Colen D, Bowen B, Stovall M, Lee A, Wang J, Drake D, Lin K, Uroskie T, Campbell CA. Reducing Infectious Complications in Implant Based Breast Reconstruction: Impact of Early Expansion and Prolonged Drain Use. Ann Plast Surg. 2016 Jun;76 Suppl 4:S312-5. doi: 10.1097/SAP.0000000000000760. PMID 26914348

DOCUMENTS (2):
  • Study Protocol (2022-11-14): https://cdn.clinicaltrials.gov/large-docs/38/NCT05846438/Prot_000.pdf
  • Informed Consent Form (2022-10-12): https://cdn.clinicaltrials.gov/large-docs/38/NCT05846438/ICF_001.pdf